CLINICAL TRIAL: NCT06313151
Title: The 2019 EULAR/ACR Classification Criteria as Predictor of Organ Damage in Systemic Lupus Erythematosus Patients
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Aliaa Abdelhameed, Assistant lecturer, Sohag University
Other Study IDs: Soh-Med-24-02-02MD
Record Dates: First submitted 2024-03-10; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: SLE, and Organ Damage Index
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to investigate if the 2019 EULAR/ACR classification criteria can be used to assess organ damage in patients with systemic lupus erythematosus (SLE) and as predictor for prognosis .

DETAILED DESCRIPTION:
The study will include 200 systemic lupus patient attending Sohag University Hospital from march 2024 to march 2025 in Rheumatology Department.

The patients included in the study will be classified as SLE patient according to 2019 ACR/EULAR classification criteria.

Inclusion criteria:

1. Patient age is above 16 years old
2. Patient is classified as SLE patient according to 2019 ACR/EULAR classification criteria
3. patient with disease duration more than 6 month.

Exclusion criteria:

1. Patient with drug-induced lupus and those with systemic sclerosis or dermatomyositis overlap syndromes .
2. patient with disease duration less than 6 month will be excluded.

Methods:

All patient will be selected randomly and undergo a complete history taking and physical examination, The data will be collected and analyzed as the following:

1. Demographic data: age, gender,sex.
2. Clinical data:

   O Age of disease onset ,disease duration, time of disease onset, organs involved , O presence of hypertension, hyperlipidemia, or diabetes, O drugs administration of hydroxychloroquine , azathioprine , cyclophosphamide pulse, cyclosporine, mycophenolate mofetil, prednisolone, and use of pulses of methylprednisolone.
3. disease activity measured by SLEDAI.

Laboratory results:

routine investigations: white cell count, hemoglobin, platelet,serum creatinine, ALT ,AST and urine analysis.

oAntinuclear antibody (ANA) by immunofluorescence and its pattern oANA profile

* Complement C3,C4.
* anticardiolipin antibody (ACA), lupus anticoagulant (LA). O Further investigation will be customized to the patient according to their clinical history and examination like abdominal ultra sound,24 hours urine protein ,glumerular filteration rate ,renal biopsy, x-ray on chest or vertebral colon, CT chest or brain, MRI brain , ECG, echo cardiography.

The organ damage assessment with the SLICC/ACR Damage Index (SDI) contains items that represent permanent, irreversible damage in a lupus patient. Items should be present for at least 6 months with the exception that manifestations such as myocardial infarction and stroke are recorded once they occur. Damage is defined for 12 organ systems: ocular (range 0-2), neuropsychiatric (0-6), renal (0-3), pulmonary (0-5), cardiovascular (0-6), peripheral vascular (0-5), gastrointestinal (0-6), musculoskeletal (0-7), skin (0-3), endocrine (diabetes) (0-1), gonadal (0-1), and malignancies (0-2). Damage over time can only be stable or increase, theoretically to a maximum of 47 points(6).

ELIGIBILITY:
Inclusion Criteria:

1. Patient age is above 16 years old
2. Patient is classified as SLE patient according to 2019 ACR/EULAR classification criteria
3. patient with disease duration more than 6 month.

Exclusion Criteria:

1. Patient with drug-induced lupus and those with systemic sclerosis or dermatomyositis overlap syndromes .
2. patient with disease duration less than 6 month will be excluded.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study will include 200 systemic lupus patient attending Sohag University Hospital from march 2024 to march 2025 in Rheumatology Department.
  The patients included in the study will be classified as SLE patient according to 2019 ACR/EULAR classification criteria.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-03-10 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
prediction organ damage in SLE by using 2019 EULAR/ACR classification criteria. | wihe in 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University, Sohag, Egypt